CLINICAL TRIAL: NCT01243047
Title: Intermittent Versus Continuous Erlotinib With Concomitant Modified 'Xelox' (q3W) in First-line Treatment of Metastatic Colorectal Cancer
Brief Title: Intermittent Versus Continuous Tarceva Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CCTU, Comprehensive Clinical Trial Unit, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COL012
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Second line treatment for metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Active Comparator): Continuous erlotinib administration (21-day cycle). Erlotinib dose given at 100mg daily
  Interventions: Drug: Chemotherapy
- Arm B (Active Comparator): Intermittent erlotinib administration (21-day cycle). Erlotinib dose given at 150mg.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Erlotinib, Oxaliplatin, Capecitabine

SUMMARY:
This is a randomized phase II study comprising of two treatment arms in patients who are previously untreated for metastatic or recurrent colorectal cancer.

DETAILED DESCRIPTION:
To evaluate two different schedules of erlotinib in combination with a modified XELOX regimen in terms of response rate

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* ECOG performance status of 0-2.
* Histological proof of adenocarcinoma of colon or rectum with evidence of metastatic disease.
* At least one unidimensionally measurable lesion with a diameter >20 mm using conventional CT or MRI scans, or > 10 mm with spiral CT
* No prior drug treatment or chemotherapy for metastatic disease.
* No prior HER2 or EGFR inhibitors. No prior Oxaliplatin in any clinical setting.
* Absolute granulocyte count > 1.5 x 109/L, platelet count > 100 x 109/L, hemoglobin level > 9.0 g/L, INR < 1.5.
* Adequate renal & hepatic functions: serum creatinine < 1.5 x upper limit of normal (ULN) or calculated creatinine clearance > 50ml/min, serum bilirubin < 1.5 x ULN, ALT < 2.5 x ULN or < 5 x ULN in case of liver metastases, albumin level > 30g/dL).
* Prior adjuvant or neoadjuvant chemotherapy for non-metastatic CRC is allowed if > 3 months has elapsed since the last dose of chemotherapy.
* Prior open surgery is allowed if > 28 days* has elapsed since the date of surgery, wound healing is satisfactory and recovery from any complications from the surgery is adequate. (*For laparoscopic surgery, > 14 days from the date of surgery).
* No serious medical conditions such as myocardial infarction within 6 months prior to entry, or any other medical conditions that might be aggravated by treatment

Exclusion Criteria:

* Prior history of any malignancies, except basal cell cancer of skin, cervical CIN.
* Treatment with radiotherapy < 30 days.
* Pregnant or lactating females
* Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study.
* Patients who have not recovered from surgery or other medical illness such as infection.
* Evidence of central nervous system disease. Patients with a history of uncontrolled seizures, central nervous disorders or psychiatric disability judged by the investigator to be clinically significant precluding informed consent or interfering with compliance for oral drug intake should be excluded from the study
* Patients lacking physical integrity of upper gastrointestinal tract or malabsorption syndrome or unable to swallow tablets.
* Prior unanticipated severe reaction to fluoropyrimidine therapy (with or without documented DPD deficiency).
* Interstitial pneumonia or extensive symptomatic fibrosis of the lungs.
* Requirement for concurrent use of the antiviral agent sorivudine (antiviral) or chemically related analogues, such as brivudine.
* Known peripheral neuropathy ≥ NCI CTC grade 1.
* Current or recent (within 10 days prior to study treatment start) use of full-dose oral anticoagulant (e.g. warfarin) or thrombolytic agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To evaluate two different schedules of erlotinib in combination with a modified XELOX regimen in terms of response rate | 3 years

SECONDARY OUTCOMES:
To evaluate two different schedules of erlotinib and modified XELOX regimen in terms of toxicity, their duration of response and effect on time to progression, progression-free survival and overall survival. | 3 years
To determine the effect of intermittent versus continuous erlotinib administration on pharmacodynamic endpoints using tumor biopsies | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Brigette Ma, MD, FRACP, Principal Investigator — Department of Clinical Oncology, The Chinese University of Hong Kong
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong